CLINICAL TRIAL: NCT05335161
Title: A New Heat Therapy Device for Home-based Leg Heating in Patients With Lower-extremity Peripheral Artery Disease: a Pilot Study
Brief Title: A New Heat Therapy Device for Home-based Leg Heating in Patients With Lower-extremity Peripheral Artery Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Aquilo Sports (Unknown)
Responsible Party: Principal Investigator, Bruno Roseguini, Associate Professor, Purdue University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-2022-375
Record Dates: First submitted 2022-04-13; First posted 2022-04-19 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication
Keywords: heat therapy; peripheral artery disease
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Hyperthermia

STUDY DESIGN:
Intervention Model Description: Six patients with PAD will be asked to complete daily (90 min/day) home-based leg HT for 12 weeks using the newly developed system. Outcomes will be measured at baseline and at 12-week follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home-based leg heat therapy (Experimental): Patients will be provided with the Aquilo heat therapy device and will be instructed on how to operate the equipment. The device will be used in accordance to the manufacturers recommendations. Patients will be asked to apply the therapy daily in the home setting for 12 week (90 min/day, 7 days/week).
  Interventions: Device: Home-based leg heat therapy

INTERVENTIONS:
Device: Home-based leg heat therapy — The Aquilo system consists of a garment that contains an inner water-circulating pad that is compressed by air bladders. The volume of air inflating the air bladders is pressure-controlled so the garment automatically adjusts to the shape and size of all legs. The touch screen console contains pre-programmed settings for ease of use. After baseline characteristics are established, patients will be provided with the Aquilo device and will be instructed on how to operate the equipment and how to rapidly remove the system if the alarm sounds or if they have any unusual feeling. Patients in both groups will also receive a logbook to record their sessions. Patients will undergo daily home-based leg HT (90 min/day, 7 days/week) for 12 weeks. Water at 42ºC will be perfused through the water-circulating garment for 90 min, with the goal of increasing skin temperature in the calf to ~37ºC.
  Other Names: Aquilo Sports

SUMMARY:
The goal of the proposed pilot study is to evaluate the feasibility of a new leg heat therapy system treatment for patients with lower extremity PAD. The new system is comprised of leg-length water circulating pads surrounded by a separate pneumatic compression outer garment that compresses the pads against the skin for efficient heat transfer. The new leg garment is easily closed with a zipper. The air chambers automatically adjust the amount of air inflation enabling use of the garment independent of patient leg size. Six patients with PAD will be asked to complete daily (90 min/day) home-based leg HT for 12 weeks using the newly developed system. The primary study outcome is the change from baseline in walking performance on the 6-minute walk test at the 12-week follow-up. Secondary outcomes include plantar flexion power, as assessed using isokinetic dynamometry, sit-to-stand muscle power and perceived quality of life.

DETAILED DESCRIPTION:
Lower-extremity PAD is a manifestation of systemic atherosclerosis associated with increased risk of cardiovascular morbidity and mortality, diminished quality of life, physical functioning and psychological well-being. In 2015, an estimated 236 million people worldwide, most between 65 and 69 years of age, were living with PAD. Home-based leg heat therapy (HT) is emerging as a potential effective and practical treatment to increase leg blood flow and improve walking performance in patients with symptomatic PAD. In the first randomized sham-controlled trial to examine the benefits of supervised leg HT in patients with symptomatic PAD (90 min, 3 days/week for 6 weeks), we demonstrated that patients assigned to the leg heating group displayed a clinically meaningful improvement in perceived physical functioning. Building upon these findings, we recently completed a NIH-sponsored randomized clinical trial to examine the safety, tolerability, and effectiveness of home-based, unsupervised leg HT (90 min, 7 days/week for 8 weeks) in 34 patients with symptomatic PAD. Patients randomized to the HT group displayed an increase in 6-minute walk from baseline of 23 meters after 8 weeks of treatment, which is clinically meaningful for PAD patients. Importantly, home-based leg HT was also found to be safe (no skin injury), well-tolerated, and patient compliance was surprisingly high (96% completion of the prescribed treatment sessions).

Heat packs, electric heating pads, and electric blankets are widely available, but have high risk of contact burns, particularly in patients with peripheral neuropathy that is commonly associated with diabetes mellitus and PAD. An assembly of individual pads is difficult to apply and skin contact is unreliable. Water-circulating pads have been found to be safer than electric devices because they provide more reliable thermostatic control. PAD patients with diffuse bilateral disease often accompanied by neuropathy need a reliable system that is simple to operate, easy to put on, covers the entirety of both lower limbs and safely provides HT while avoiding skin injury. Currently, there is no commercially-available HT system for home-based therapy in elderly individuals, despite the documented benefits associated with repeated HT. To address this unmet clinical need, Aquilo Sports is developing a system that will monitor skin temperature and have an integrated shut-off feature to prevent skin burns, and record treatment sessions to confirm patient compliance. The system has undergone extensive independent validation testing and has been widely adopted by professional athletes. The garment is easily closed with a zipper and auto-adjusts pneumatically to different leg sizes.

Our objective is to establish evidence to support the safety and feasibility of the redeveloped Aquilo system during repeated home-based treatment in patients with PAD. Our approach to testing our hypothesis will be to ask 6 patients with PAD to undergo daily home-based leg HT (90 min/day, 7 days/week) for 12 weeks. The length of the intervention (12 weeks) was selected as it is similar to: 1) the duration of previous studies with other HT modalities showing beneficial effects in patients with PAD, 2) the recommended minimal duration of exercise training interventions, the gold standard treatment for PAD.

The primary study outcome is the change from baseline in walking performance on the 6-minute walk test at the 12-week follow-up. Secondary outcomes include plantar flexion power, as assessed using isokinetic dynamometry, sit-to-stand muscle power and perceived quality of life.The study coordinator will call patients weekly to record the occurrence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 60 years or older
* Resting ankle-brachial index (ABI) of 0.9 or less in at least one leg.
* Individuals with a resting ABI between 0.91 and 1.00 at baseline will be eligible if their ABI drops by 20% or greater following a heel-rise test.

Exclusion Criteria:

* Critical limb ischemia (ischemic rest pain or ischemia-related, non-healing wounds or tissue loss)
* Prior amputation
* Exercise tolerance limited by factors other than leg pain (e.g. angina, arthritis, severe lung disease, etc).
* Recent (<3 months) lower-extremity revascularization or orthopedic surgery
* Use of walking aid other than a cane
* Active cancer
* Chronic kidney disease (eGFR <30 by MDRD or Mayo or Cockcroft-Gault formula)
* Unable to fit into water-circulating trousers
* A Mini-Mental Status Examination score <23
* Impaired thermal sensation in the leg
* Age lower than 60 yrs

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Device feasibility, safety, and usability were evaluated in an open-label, single-arm pilot study performed at Purdue University in West Lafayette, Indiana. Participants were provided the prototype HT device and were asked to apply the therapy daily (90 minutes, 7 days/week) for 12 weeks. The first participant was enrolled on May 30, 2023. The final follow-up occurred on February 7, 2024.
Pre-assignment Details: Participants attended two baseline laboratory visits. No run-in or wash-out period was used, and no participants were excluded between enrollment and assignment.
Period: Overall Study
Arm/Group | Home-based Leg Heat Therapy
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Home-based Leg Heat Therapy
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Six-minute Walk Distance
Description: Participants will receive standardized instructions and will be asked to walk the greatest distance possible by walking back and forth along a 100-ft corridor for 6 min.
Time Frame: Baseline to 12-week follow-up
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Home-based Leg Heat Therapy
Number analyzed (Participants) | 6
Meters | 32.3 (39)

2. Secondary Outcome: Change in Walking Impairment Questionnaire Score
Description: This disease-specific questionnaire assess the ability of patients with PAD to walk defined distances and speeds and to climb stairs, with scores ranging from 0 to 100. Higher scores indicate better walking ability (i.e., better outcome). Lower scores indicate greater walking impairment (i.e., worse outcome)
Time Frame: Baseline to 12-week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Leg Heat Therapy
Number analyzed (Participants) | 6
score on a scale | 11.08 (16.79)

3. Secondary Outcome: Device Usability Using the System Usability Scale
Description: Scores range from 0 to 100; > 70 represents acceptable usability.
Time Frame: Baseline to 12-week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Leg Heat Therapy
Number analyzed (Participants) | 6
score on a scale | 49 (11.98)

4. Secondary Outcome: Change in Triceps Surae Peak Torque
Description: Torque assessments of the plantar flexors will be performed using an isokinetic dynamometer. Participants will be asked to perform 3 maximal contractions.
Time Frame: Baseline to 12-week follow-up
Measure: Mean (Standard Deviation); unit: Nm
Arm/Group | Home-based Leg Heat Therapy
Number analyzed (Participants) | 6
Nm | 4.49 (6.33)

5. Secondary Outcome: Change in the Five Times Sit to Stand Test
Description: Participants were asked to sit in a chair with arms folded across their chest and stand five times consecutively as quickly as possible. The time it took to complete five chair rises was measured.
Time Frame: Baseline to 12-week follow-up
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Home-based Leg Heat Therapy
Number analyzed (Participants) | 6
Seconds | -1.93 (2.55)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Arm/Group | Home-based Leg Heat Therapy
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT05335161/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT05335161/ICF_001.pdf